CLINICAL TRIAL: NCT07154849
Title: Comparative Study Between the Efficacy of Intravenous Hydrocortisone and Intravenous Dexmedetomidine for Prevention of Postoperative Shivering After General Anaesthesia for Abdominal Surgeries
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, maha sadek El Derh, assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU MS581 /2024
Record Dates: First submitted 2025-08-13; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-09

CONDITIONS: Shivering
MeSH Terms: interventions — Hydrocortisone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A:(Hydrocortisone group) (Active Comparator): • Group A: : received 2mg/kg.
  Interventions: Drug: Hydrocortisone
- Group B: (Dexmedetomidine group) (Active Comparator): • Group B: : received 1 µg/kg.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Hydrocortisone — received 2mg/kg.
  Arms: Group A:(Hydrocortisone group)
Drug: Dexmedetomidine — received 1 µg/kg
  Arms: Group B: (Dexmedetomidine group)

SUMMARY:
The aim and purpose of this study is to compare the efficacy of intravenous hydrocortisone and intravenous dexmedetomidine for prevention and treatment of postoperative shivering after general anesthesia for abdominal surgeries.

DETAILED DESCRIPTION:
* . Type of Study: Randomized controlled clinical trial.
* Study Settings: Ain Shams University hospitals, Cairo, Egypt.
* Study Population: patients undergoing abdominal open surgeries with general anesthesia.
* Inclusion Criteria:
* ASA I or ASA II patients Scheduled for abdominal surgery under general anaesthesia.
* Age between18-65 years.
* Procedure duration ≤ 120 minutes.
* Exclusion Criteria:
* Patients with known neurologic and psychiatric illness.
* Uncontrolled diabetic patients.
* Patients on long term steroid therapy.
* Allergy to any of the drugs used in the study.
* Pregnancy and lactation.
* Hypo or hyperthyroidism.
* Sampling Method: Simple randomization
* Standard care Standard care for all patients undergoing this study will be done by senior staff expert members of Ain-Shams University Anesthesia department and will be monitored by supervisors.
* Study Procedures:
* Preoperative settings:

All patients will be assessed preoperatively by careful history taking, full physical examination, and laboratory evaluation. An informed written consent will be taken from every patient just before the surgery.

• Intraoperative and postoperative settings:

Patients will be divided into two groups:

* Group A: (HYDROCORTISONE group): will receive 2mg/kg .
* Group B: (Dexmedetomidine group): will receive 1 µg/kg . On arrival to the operating room, routine monitors will be applied, including a blood pressure cuff, electrocardiogram, pulse oximeter, and capnogram. core temperature will be measured using temperature probe to determine baseline values. An intravenous ringer infusion will be started. Pre oxygenation will be done with 100% oxygen on 6L\m for 3 minutes. Anesthesia will be induced with propofol 2 mg/kg, fentanyl 2 mic\kg and atracurium 0.5 mg/kg. After endotracheal intubation, anesthesia will be maintained with 1.2-1.5% isoflurane. Mechanical ventilation will be adjusted to maintain end-tidal carbon dioxide tension at 30-35 mmHg Patients will be covered with surgical drapes. Supplemental doses of atracurium will be given every 20 minutes to maintain muscle relaxation during surgery.

Approximately 30 minutes before the anticipated completion of surgery, the study drugs will be given to the two groups.

Ephedrine (10 mg IV bolus) will be given for hypotension (systolic blood pressure < 80 mmHg) and atropine (0.5 mg IV bolus) will be given for bradycardia (HR < 50 BPM).

At the end of surgery, extubation will be done and patients will be transferred to the post-anaesthesia care unit (PACU), for further monitoring.

• Postoperative settings: Patients will be transferred to the post-anaesthesia care unit (PACU) and will be put under observation for 30 minutes.

• Measurements: Baseline core temperature (pre-induction) will be taken as the first measurement in the operating room. Heart rate and non-invasive blood pressure readings will be recorded.

Core temperature will be measured directly after endotracheal intubation and every 15 minutes during the operation. Upon transferal of the patient to the post-anesthesia care unit (PACU), core temperature will be measured and shivering will be graded from (0-3) according to the shivering scale validated by Crossley and Mahajan as follows: 0 = no shivering, 1 = mild fasciculation of the face or neck, 2 = visible tremor involving more than one muscle group, 3 = gross muscular activity involving the entire body.

• Primary outcome: To compare the efficacy of hydrocortisone and dexmedetomidine in reducing shivering post operatively.

• Secondary outcomes: Measurement of the hemodynamic changes if present.

ELIGIBILITY:
Inclusion Criteria: any patient undergoing abdominal surgery ASAI or II.

-

Exclusion Criteria:

* Patients with known neurologic and psychiatric illness.
* Uncontrolled diabetic patients.
* Patients on long term steroid therapy.
* Allergy to any of the drugs used in the study.
* Pregnancy and lactation.
* Hypo or hyperthyroidism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants with body respond to decrease in body temperature by shivering | 30 minutes
  In this study it was targeted to assess the efficacy of hydrocortisone and dexmedetomidine in reducing shivering that occur post operatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt